CLINICAL TRIAL: NCT04041596
Title: A Phase IV, Single-center Study of the Benefits of the Advanced Bionics Naída CI Q90 Acoustic Earhook in Adults Cochlear Implant Recipients.
Brief Title: Degree of Benefit From Low-Frequency Acoustic Amplification Using the Advanced Bionics Acoustic Earhook
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to a lack of enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01276
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Cochlear Implant; Cochlear Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Advanced Bionics' Acoustic Earhook — designed to deliver acoustic amplification through the modular attachment of the Naída CI Q90 AcoustiEarhook, while also delivering electrical stimulation along the full range of the implanted Advanced Bionics electrode.

SUMMARY:
The primary objective of this study is to obtain a greater understanding of the range in benefit from acoustic amplification combined with electric stimulation in cochlear implant recipients with low-frequency hearing who do not currently use the commercially approved Advanced Bionics Acoustic Earhook. The aims of this study are to 1) obtain subjective sound quality judgements of recorded speech and music samples, 2) assess vocal emotion perception, and 3) evaluate post-operative speech perception and sound field detection thresholds in CI recipients both with and without use of the acoustic ear hook.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Implanted with an Advanced Bionics Advanced Bionics HiRes Ultra, 90K, or CII implant, and using a Naída Q90 sound processor
* 18 years of age or older with post-lingual hearing loss
* Aided open-set speech recognition scores greater than 30% correct in quiet in the ear to be tested
* Unaided low frequency audiometric hearing thresholds of 90 dB HL or better at .125, .25, and .5 kHz
* Participants must have a working understanding of and ability to verbalize in English as the evaluation measures are available exclusively in English
* Willingness to use an acoustic component with their ear-level sound processor postoperatively for the duration of the study
* Willingness to participate in all scheduled procedures outlined in the protocol

Exclusion Criteria:

* Exclusive use of a body worn external sound processor
* Deafness due to central auditory lesion or cochlear nerve deficiency, diagnosis of auditory neuropathy/dys-synchrony in either the implanted or the contralateral ear
* Postoperative unaided low frequency audiometric hearing thresholds in the implanted ear exceeding 90 dB HL at any frequency from 125 - 500 Hz.
* Presence of other conditions that could affect performance on outcome measures or otherwise confound or interfere with study participation or outcomes measures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Change in Speech recognition testing, with and without acoustic earhook | 3 Months, 6 Months, 12 Months
  5-alternative identification task to measure vocal emotion recognition (Toronto Emotional Speech Test (TESS) at initial fitting, and 3, 6, and 12 months after fitting
Change in Sound quality judgements, with and without acoustic earhook | 3 Months, 6 Months, 12 Months
  Ratings of sound quality (Judgement of Sound Quality {JSQ} test) of speech and music samples at initial fitting, and 3, 6, and 12 months after fitting
Change in Vocal emotion perception task, with and without acoustic earhook | 3 Months, 6 Months, 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Susan Waltzman, MD, Principal Investigator — New York Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No